CLINICAL TRIAL: NCT04226742
Title: Evaluation of the Crowd-Powered Web Platform for Accumulative Depression and Anxiety Plans and Treatment (ADAPT)
Brief Title: Evaluation of a Crowd-Powered Web Platform for Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mental Health America (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Stephen Matthew Schueller, Assistant Proffessor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS#2019-4901, HS#2020-6071; 1R34MH113616-01A1 (NIH)
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either the treatment condition (ADAPT platform, iCBT platform comprised of didactic and interactive content), or a control condition (iCBT comparison platform comprised only of didactic content).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of which condition they have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants randomly assigned to this condition will receive the ADAPT platform (treatment) for a treatment period of 8 weeks.
  Interventions: Behavioral: ADAPT Platform (Treatment)
- Control (Active Comparator): Participants randomly assigned to this condition will receive a similar self-guided platform (control) for a treatment period of 8 weeks.
  Interventions: Behavioral: ADAPT Comparison (Control)

INTERVENTIONS:
Behavioral: ADAPT Platform (Treatment) — The ADAPT platform consists of 2 modules based on evidence-based strategies from cognitive-behavioral therapy including cognitive restructuring and behavioral experiments. The platform includes didactic material, interactive tools, and crowd-features. Crowd-features are present to increase personal relevance of content and to promote engagement with the ADAPT platform through accountability. Crowd-features include requesting, responding, and exemplars.
  Arms: Treatment
Behavioral: ADAPT Comparison (Control) — The control platform is a self-guided version of the ADAPT platform that includes no crowd-features. As such it will include only didactic material on cognitive restructuring and behavioral experiments and interactive tools.
  Arms: Control

SUMMARY:
100 participants will be enrolled in a two-armed randomized controlled trial of the Accumulated Depression and Anxiety Plans and Treatments (ADAPT) platform which integrates internet Cognitive Behavioral Therapy (iCBT) to determine impact on symptoms of depression and anxiety. This trial will pilot the effectiveness of the ADAPT platform, and evaluate the extent to which the ADAPT platform engages putative targets of personal relevance, skills use, and skills mastery.

DETAILED DESCRIPTION:
The investigators will enroll 100 participants in a two-armed randomized controlled trial of the ADAPT platform (iCBT). Participants will be randomly assigned to receive either the ADAPT platform (treatment) or a similar self-guided platform (control) that contains the didactic material (learning) but lacks the ADAPT platforms "crowd" features. Participants will use their assigned platform for a treatment period of 8 weeks. Participants will receive trial assessments at baseline, week 4, and week 8 (post-treatment). Follow-up evaluations will occur at 16 weeks to evaluate maintenance of gains. This pilot effectiveness trial aims to determine the impact on symptoms of depression and anxiety and whether the platform engages the putative targets of personal relevance, relationship, resulting in increased skills mastery and skills use.

ELIGIBILITY:
Inclusion Criteria:

* 1) Completion of the Mental Health America Screening to Supports (MHA S2S) or significant mood and anxiety symptoms as defined by an accepted cut-off on a validated measure the Depression Anxiety and Stress Scale (DASS). The accepted cut-off is scores greater than 22;
* 2) able to speak and read English;
* 3) at least 18 years of age.

Exclusion Criteria:

* 1) severe suicidality (has ideation, plan, and intent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Schueller, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will be deposited into the NIH data repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available immediately following publication, no end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Dear BF, Titov N, Schwencke G, Andrews G, Johnston L, Craske MG, McEvoy P. An open trial of a brief transdiagnostic internet treatment for anxiety and depression. Behav Res Ther. 2011 Dec;49(12):830-7. doi: 10.1016/j.brat.2011.09.007. Epub 2011 Sep 28. PMID 21993153
- [Background] Titov N, Dear BF, Schwencke G, Andrews G, Johnston L, Craske MG, McEvoy P. Transdiagnostic internet treatment for anxiety and depression: a randomised controlled trial. Behav Res Ther. 2011 Aug;49(8):441-52. doi: 10.1016/j.brat.2011.03.007. Epub 2011 Apr 3. PMID 21679925
- [Background] van Ballegooijen W, Cuijpers P, van Straten A, Karyotaki E, Andersson G, Smit JH, Riper H. Adherence to Internet-based and face-to-face cognitive behavioural therapy for depression: a meta-analysis. PLoS One. 2014 Jul 16;9(7):e100674. doi: 10.1371/journal.pone.0100674. eCollection 2014. PMID 25029507
- [Background] Schueller SM, Mohr DC. Initial Field Trial of a Coach-Supported Web-Based Depression Treatment. Int Conf Pervasive Comput Technol Healthc. 2015 Aug;2015:10.4108/icst.pervasivehealth.2015.260115. doi: 10.4108/icst.pervasivehealth.2015.260115. Epub 2015 Aug 3. PMID 26640741
- [Background] Munoz RF. Using evidence-based internet interventions to reduce health disparities worldwide. J Med Internet Res. 2010 Dec 17;12(5):e60. doi: 10.2196/jmir.1463. PMID 21169162
- [Background] Munoz RF, Aguilera A, Schueller SM, Leykin Y, Perez-Stable EJ. From online randomized controlled trials to participant preference studies: morphing the San Francisco Stop Smoking site into a worldwide smoking cessation resource. J Med Internet Res. 2012 Jun 27;14(3):e64. doi: 10.2196/jmir.1852. PMID 22739225
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Lovibond, S. H., & Lovibond, P. F. (1993). Manual for the Depression Anxiety Stress Scales (DASS). Psychology Foundation Monograph, University of New South Wales.
- [Background] Muñoz, R. F., Bunge, E. L., Chen, K., Schueller, S. M., Bravin, J. I., Shaughnessy, E. A., & Pérez- Stable, E. J. (2015). Massive open online interventions: A novel model for delivering behavioral-health services worldwide. Clinical Psychological Science. Advanced Online Publication. http://doi.org/10.1177/2167702615583840
- [Background] MacArthur Foundation's Initiative (2004). The Macarthur initiative on depression and primary care at Dartmouth and Duke: Depression management toolkit. Hanover, NH: Dartmouth.
- [Background] First, M. B., Williams, J. B. W., Karg, R. S., & Spitzer, R. L. (2015). Structured clinical interview for DSM-5 disorders, clinician version (SCID-5-CV). Arlington, VA: American Psychiatric Association.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Gorka SM, Lieberman L, Klumpp H, Kinney KL, Kennedy AE, Ajilore O, Francis J, Duffecy J, Craske MG, Nathan J, Langenecker S, Shankman SA, Phan KL. Reactivity to unpredictable threat as a treatment target for fear-based anxiety disorders. Psychol Med. 2017 Oct;47(14):2450-2460. doi: 10.1017/S0033291717000964. Epub 2017 Apr 24. PMID 28436351
- [Background] Gorka SM, Burkhouse KL, Afshar K, Phan KL. Error-related brain activity and internalizing disorder symptom dimensions in depression and anxiety. Depress Anxiety. 2017 Nov;34(11):985-995. doi: 10.1002/da.22648. Epub 2017 Sep 20. PMID 28940987
- [Background] Burkhouse KL, Gorka SM, Afshar K, Phan KL. Neural reactivity to reward and internalizing symptom dimensions. J Affect Disord. 2017 Aug 1;217:73-79. doi: 10.1016/j.jad.2017.03.061. Epub 2017 Mar 29. PMID 28391111
- [Background] Duffecy, J., Cai, X., & Mohr, D. C. (2013). Supportive accountability: Measurement of a framework for adherence to behavioral intervention technologies. International Society for Research on Internet Interventions, Chicago, IL.
- [Background] Miner AS, Schueller SM, Lattie EG, Mohr DC. Creation and validation of the Cognitive and Behavioral Response to Stress Scale in a depression trial. Psychiatry Res. 2015 Dec 30;230(3):819-25. doi: 10.1016/j.psychres.2015.10.033. Epub 2015 Oct 30. PMID 26553147
- [Background] Chesney MA, Neilands TB, Chambers DB, Taylor JM, Folkman S. A validity and reliability study of the coping self-efficacy scale. Br J Health Psychol. 2006 Sep;11(Pt 3):421-37. doi: 10.1348/135910705X53155. PMID 16870053
- [Background] Hahn EA, Devellis RF, Bode RK, Garcia SF, Castel LD, Eisen SV, Bosworth HB, Heinemann AW, Rothrock N, Cella D; PROMIS Cooperative Group. Measuring social health in the patient-reported outcomes measurement information system (PROMIS): item bank development and testing. Qual Life Res. 2010 Sep;19(7):1035-44. doi: 10.1007/s11136-010-9654-0. Epub 2010 Apr 25. PMID 20419503
- [Background] Hollandare F, Johnsson S, Randestad M, Tillfors M, Carlbring P, Andersson G, Engstrom I. Randomized trial of Internet-based relapse prevention for partially remitted depression. Acta Psychiatr Scand. 2011 Oct;124(4):285-94. doi: 10.1111/j.1600-0447.2011.01698.x. Epub 2011 Mar 14. PMID 21401534
- [Background] Titov N, Dear BF, Johnston L, Lorian C, Zou J, Wootton B, Spence J, McEvoy PM, Rapee RM. Improving adherence and clinical outcomes in self-guided internet treatment for anxiety and depression: randomised controlled trial. PLoS One. 2013 Jul 3;8(7):e62873. doi: 10.1371/journal.pone.0062873. Print 2013. PMID 23843932
- [Background] Kelders SM, Bohlmeijer ET, Pots WT, van Gemert-Pijnen JE. Comparing human and automated support for depression: Fractional factorial randomized controlled trial. Behav Res Ther. 2015 Sep;72:72-80. doi: 10.1016/j.brat.2015.06.014. Epub 2015 Jul 6. PMID 26196078
- [Background] Smith P, Scott R, Eshkevari E, Jatta F, Leigh E, Harris V, Robinson A, Abeles P, Proudfoot J, Verduyn C, Yule W. Computerised CBT for depressed adolescents: Randomised controlled trial. Behav Res Ther. 2015 Oct;73:104-10. doi: 10.1016/j.brat.2015.07.009. Epub 2015 Jul 21. PMID 26301756
- [Background] Johnston L, Titov N, Andrews G, Dear BF, Spence J. Comorbidity and internet-delivered transdiagnostic cognitive behavioural therapy for anxiety disorders. Cogn Behav Ther. 2013;42(3):180-92. doi: 10.1080/16506073.2012.753108. Epub 2013 Mar 4. PMID 23458319
- [Background] Titov N, Dear BF, Staples LG, Bennett-Levy J, Klein B, Rapee RM, Shann C, Richards D, Andersson G, Ritterband L, Purtell C, Bezuidenhout G, Johnston L, Nielssen OB. MindSpot Clinic: An Accessible, Efficient, and Effective Online Treatment Service for Anxiety and Depression. Psychiatr Serv. 2015 Oct;66(10):1043-50. doi: 10.1176/appi.ps.201400477. Epub 2015 Jul 1. PMID 26130001
- [Background] Kirkpatrick T, Manoukian L, Dear BF, Johnston L, Titov N. A feasibility open trial of internet-delivered cognitive-behavioural therapy (iCBT) among consumers of a non-governmental mental health organisation with anxiety. PeerJ. 2013 Nov 28;1:e210. doi: 10.7717/peerj.210. eCollection 2013. PMID 24349897
- [Background] van Mierlo T. The 1% rule in four digital health social networks: an observational study. J Med Internet Res. 2014 Feb 4;16(2):e33. doi: 10.2196/jmir.2966. PMID 24496109
- [Background] Christensen H, Griffiths K, Groves C, Korten A. Free range users and one hit wonders: community users of an Internet-based cognitive behaviour therapy program. Aust N Z J Psychiatry. 2006 Jan;40(1):59-62. doi: 10.1080/j.1440-1614.2006.01743.x. PMID 16403040
- [Background] Eysenbach G. The law of attrition. J Med Internet Res. 2005 Mar 31;7(1):e11. doi: 10.2196/jmir.7.1.e11. PMID 15829473
- [Background] Mohr DC, Tomasino KN, Lattie EG, Palac HL, Kwasny MJ, Weingardt K, Karr CJ, Kaiser SM, Rossom RC, Bardsley LR, Caccamo L, Stiles-Shields C, Schueller SM. IntelliCare: An Eclectic, Skills-Based App Suite for the Treatment of Depression and Anxiety. J Med Internet Res. 2017 Jan 5;19(1):e10. doi: 10.2196/jmir.6645. PMID 28057609
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] Braithwaite SR, Giraud-Carrier C, West J, Barnes MD, Hanson CL. Validating Machine Learning Algorithms for Twitter Data Against Established Measures of Suicidality. JMIR Ment Health. 2016 May 16;3(2):e21. doi: 10.2196/mental.4822. PMID 27185366
- [Background] O'Dea, B., Wan, S., Batterham, P. J., Calear, A. L., Paris, C., & Christensen, H. (2015). Detecting suicidality on Twitter. Internet Interventions, 2(2), 183-188. http://dx.doi.org/10.1016/j.invent.2015.03.005
- [Background] Nguyen, T., O'Dea, B., Larsen, M., Phung, D., Venkatesh, S., & Christensen, H. (2015, November). Differentiating sub-groups of online depression-related communities using textual cues. In International Conference on Web Information Systems Engineering (pp. 216-224). Springer International Publishing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Mental Health America screening website between Feburary 2021 and September 2021. The first participant was enrolled on February 18, 2021 and the last participant was enrolled on September September 3, 2021.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 56 | 51
Completed | 35 | 35
Not Completed | 21 | 16
Not completed — Lost to Follow-up | 16 | 13
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 56 | 51 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.41 (11.41) | 34.57 (13.39) | 33.92 (12.34)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 22 | 19 | 41
  Non-Binary | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 21
  Not Hispanic or Latino | 48 | 37 | 85
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 36 | 32 | 68
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 1 | 5 | 6
Depression Anxiety Stress Scale (DASS) [Mean (Standard Deviation); unit: scores on a scale] — DASS total score with scores ranging from 21 to 84 with lower values (21 = lowest) indicating lower levels of depression, anxiety, and stress and higher values (84 = highest) indicating higher levels of depression, anxiety, and stress.
  scores on a scale | 65.7 (23.8) | 63.2 (24.3) | 64.51 (24.06)

OUTCOME MEASURES:

1. Primary Outcome: Depression Scores at Week 16
Description: The primary outcome of symptoms of depression will be measured with the self-report depression subscale of the Depression Anxiety Stress Scale (DASS). The subscale for depression ranges from 7 to 28 with lower values (lowest value = 7) indicating lower levels of depression and higher values (highest value = 28) indicating higher levels of depression.
Time Frame: Absolute scores at Week 16
Population: Data was analyzed using an intent-to-treat analysis including all participants who provided baseline data entered into a mixed models analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 15.7 (12.9) | 15.7 (10.3)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.79, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = 0.58, 95% CI 2-sided [-3.71 to 4.88]

2. Primary Outcome: Anxiety Scores at 16 Weeks
Description: The primary outcome of symptoms of anxiety will be measured with the self-report anxiety subscale of the Depression Anxiety Stress Scale (DASS). The subscale for anxiety ranges from 7 to 28 with lower values (lowest value = 7) indicating lower levels of anxiety and higher values (highest value = 28) indicating higher levels of anxiety.
Time Frame: Absolute scores at Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 12.4 (10.8) | 11.0 (9.77)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .61, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = 0.90, 95% CI 2-sided [-2.52 to 4.32]

3. Secondary Outcome: Cognitive and Behavioral Skills Scores at 16 Weeks
Description: A secondary outcome is the Frequency of Actions and Thoughts (FATS), which assesses the use of cognitive and behavioral skills. Total scores indicate the average of each item rating and range from 0-4. Lower scores indicate less frequent use of cognitive and behavioral skills and higher scores indicate more frequent use of cognitive and behavioral skills.
Time Frame: Absolute scores at Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 2.03 (0.84) | 1.78 (0.90)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.088, Mixed Models Analysis — Significance threshold of alpha = 0.05; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.05 to 0.68]

4. Secondary Outcome: Self-efficacy Scores at 16 Weeks
Description: A secondary outcome is the Coping Self-Efficacy (CSE), which produces a single score that ranges from 0-260 with lower scores representing lower coping self-efficacy and higher scores indicating higher coping self-efficacy.
Time Frame: Absolute scores at Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 56 | 51
score on a scale | 134.0 (58.6) | 124.0 (57.8)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.142, Mixed Models Analysis — Threshold for statistical significance of alpha = 0.05; Mean Difference (Final Values) = 13.68, 95% CI 2-sided [-4.62 to 31.99]

5. Secondary Outcome: Accountability Scores at 16 Weeks
Description: A secondary outcome is the Supportive Accountability Questionnaire (SAQ), which produces a single score than ranges from 7-91. Data reported are the SAQ total scores with lower levels indicating less supportive accountability and higher values indicating greater supportive accountability.
Time Frame: Absolute scores at Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
score on a scale | 75.1 (23.3) | 74.7 (22.0)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.109, Mixed Models Analysis — Threshold for statistical significance of alpha = .05; Mean Difference (Final Values) = -6.87, 95% CI 2-sided [-15.28 to 1.54]

6. Secondary Outcome: Social Functioning Scores at 16 Weeks
Description: Functioning will be assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities Scale which produces T-scores that have a mean of 50 and a standard deviation of 10. Lower scores indicate lower participation in social roles and activities and higher scores indicate higher participation in social roles and activities.
Time Frame: Absolute scores at Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 35
T-score | 78.4 (14.2) | 79.3 (16.0)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.736, Mixed Models Analysis; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-6.92 to 4.89]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/51
Other Adverse Events (participants affected / at risk) | 0/56 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04226742/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04226742/SAP_001.pdf
  • Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT04226742/ICF_002.pdf